CLINICAL TRIAL: NCT05914948
Title: Minimally Invasive Electrical Stimulation Of The Nerve Hypoglossal for the Treatment of Obstructive Sleep Apnea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capri Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CAP 001
Record Dates: First submitted 2023-06-09; First posted 2023-06-22 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; hypopnea syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Subjects meeting study eligibility criteria will be implanted with a Medtronic 8-contact Vectris subcompact or compact electrode.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Subjects implanted with a Medtronic 8-contact Vectris subcompact or compact electrode. (Other): Subjects meeting study eligibility criteria will be implanted with a Medtronic 8-contact Vectris subcompact or compact electrode.
  Interventions: Device: Medtronic 8-contact Vectris subcompact or compact electrode.

INTERVENTIONS:
Device: Medtronic 8-contact Vectris subcompact or compact electrode. — Subjects meeting study eligibility criteria will be implanted with a Medtronic 8-contact Vectris subcompact or compact electrode.

SUMMARY:
Minimally invasive electrical stimulation of the nerve hypoglossal for the treatment of obstructive sleep apnea.

To demonstrate the correct stimulation of the medial branches of the hypoglossal nerve and tongue protrusion using a minimally invasive implantation technique in patients with OSA.

DETAILED DESCRIPTION:
Study title: Minimally invasive electrical stimulation of the nerve hypoglossal for treatment for obstructive sleep apnea.

Study device: Medtronic 8-contact Vectris subcompact or compact electrode.

Study design: This is an initial feasibility study that seeks to determine the safety and effectiveness of a minimally invasive technique to implant a hypoglossal nerve stimulation electrode in patients with obstructive sleep apnea.

Subjects meeting study eligibility criteria will be implanted with a Medtronic 8-contact Vectris subcompact or compact electrode.

In the follow-up visits, quality of life and sleepiness scales (Epworth) will be performed, and on days 4 and 7 a control polysomnography. All results will be compared with the baseline data obtained at the start of the study.

Study Size: Up to 30 subjects may be enrolled to achieve a number of implanted subjects between 10 to 20.

Study Duration: Total expected duration per subject is approximately 10 days. The study is estimated to take 6 months.

Objective of the study: The main objective is to evaluate the safety and effectiveness of a minimally invasive technique to implant a hypoglossal nerve stimulation electrode in patients with obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

1. Age >22 and <75 years
2. Moderate or severe apnea (Apnea-Hypopnea Index, AHI, between 1550 per hour and <25% of central apneas)
3. Failure of continuous positive airway pressure (CPAP) therapy defined as the inability to eliminate obstructive sleep apnea and hypopnea syndrome (OSAHS) corresponding to an AHI greater than 20/h despite the use of CPAP.
4. No tolerance to CPAP:

   to. Inability to use CPAP (more than 5 nights a week; more than 4 hours a night).

   b. Unwillingness to use CPAP (for example, a patient returns the CPAP system after trying to use it).
5. Patients willing and able to give their informed consent.
6. Willing and able to have a pacing system temporarily implanted, and use the patient programmer to activate the stimulation.
7. Willing and able to return for all follow-up visits and sleep studies and able to fill out questionnaires.

Exclusion Criteria:

1. Body mass index (BMI) >32 kg/m.
2. Central or mixed apneas > or = 25%.
3. Patients who are pregnant or planning to become pregnant.
4. Presence of a complete collapse at the level of the palate corroborated by drug-induced endoscopy (DISE).
5. Surgical resection or radiation therapy for cancer or congenital malformations of the larynx, tongue, or throat.
6. Significant comorbidities that make the patient unable or inappropriate to participate in the trial.
7. Patients with a history of lack of response to electrical stimulation of the hypoglossal nerve.
8. Patients with the presence of other implantable electrical devices such as:

spinal cord stimulator, pacemaker, cochlear implant, peripheral nerve stimulator, etc.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | 6 months
  Demonstrate an AHI reduction from baseline of 50% and an AHI less than 20 on follow-up polysomnography
Oxygen Desaturation Index (ODI) | 6 months
  Demonstrate at least a 25% reduction in the ODI from the initial value.
Security | 6 months
  The primary safety objective is to assess the incidence of events Adverse events related to the device and the insertion technique

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica de Otorrinolaringología de Antioquia (ORLANT), Medellín, Antioquia, Colombia